CLINICAL TRIAL: NCT05805657
Title: Implementing and Sustaining a Transdiagnostic Sleep and Circadian Treatment to Improve Severe Mental Illness Outcomes in Community Mental Health Part 2: Train-the-Trainer
Brief Title: Implementing and Sustaining a Sleep Treatment to Improve Community Mental Health Part 2: Train-the-Trainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH120147_P2; R01MH120147 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-04-10 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Sleep Disorder; Circadian Dysregulation
MeSH Terms: conditions — Sleep Wake Disorders; Chronobiology Disorders | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: CMHC sites will be cluster randomized to either Standard TranS-C or Adapted TranS-C. Then within each CMHC site, patients will be randomized to either TranS-C or to Usual Care followed by Delayed Treatment (UC-DT).
Who Masked: Outcomes Assessor
Masking Description: The assessment team will be blind to group allocation at post-treatment and six-month follow-up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard TranS-C (Experimental): Standard TranS-C is modularized and delivered across eight 50-minute, weekly, individual sessions. It is comprised of 4 cross-cutting interventions featured in every session; 4 core modules that apply to the vast majority of patients; and 7 optional modules used less commonly, depending on the presentation.
  Interventions: Behavioral: Standard Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C)
- Adapted TranS-C (Experimental): The process for developing Adapted TranS-C has been iterative and grounded in theory, data and stakeholder feedback. The core elements of the evidence-based theory of change underpinning TranS-C have been retained. Adapted TranS-C is delivered in four 20-minute, weekly, individual sessions.
  Interventions: Behavioral: Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C)
- UC-DT (Active Comparator): Usual Care Delayed Treatment. Usual care in the partner CMHCs starts with a case manager who co-ordinates care and refers each client for a medication review and to various rehabilitation programs (e.g., health care, housing, nutrition, finding a job, peer monitoring).
  Interventions: Other: Usual Care Delayed Treatment

INTERVENTIONS:
Behavioral: Standard Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) — TranS-C is a psychosocial treatment designed to improve sleep and circadian functioning. It is a modular, psychosocial, skills-based approach. In this study, two version of TranS-C will be tested: Standard and Adapted.
  Arms: Standard TranS-C
Behavioral: Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) — The Adapted version was derived from Standard TranS-C. It was developed to improve the fit of the treatment with the CMHC context.
  Arms: Adapted TranS-C
Other: Usual Care Delayed Treatment — Usual care in the partner CMHCs typically starts with a case manager who co-ordinates care and refers each client for a medication review and to various rehabilitation programs (e.g., health care, housing, nutrition, finding a job, peer monitoring).
  Arms: UC-DT

SUMMARY:
The train-the-trainer (TTT) approach is a promising method of sustaining training efforts in community mental health centers (CMHCs). This study will test the implementation and effectiveness outcomes of a sleep treatment delivered by CMHC providers who are trained and supervised within CMHCs via TTT. The investigators will test two versions of the sleep treatment, a "Standard" version and an "Adapted" version that has been adapted using theory, data and stakeholder inputs to improve the fit for SMI patients treated in community mental health centers.

DETAILED DESCRIPTION:
There are significant barriers to widespread implementation and sustainment of evidence-based psychological treatments (EBPTs) in community mental health centers (CMHCs), including insufficient time and funding, shortage of trainers and consultants, and staff turnover. The investigators propose to evaluate one possible solution, the train-the-trainer (TTT) approach, in the context of a transdiagnostic EBPT for sleep and circadian dysfunction-the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C)- for serious mental illness (SMI) in CMHCs. This entry describes the Train-the-Trainer Phase, the second of a three-phase hybrid type 2 effectiveness-implementation trial conducted to test TranS-C in CMHCs.

TTT is a training structure with multiple levels, called "Generations." First, external expert trainers train an initial cohort of providers in a specific EBPT ("Generation 1 providers"). Next, Generation 1 providers are offered additional training in how to train others in the EBPT and become "local trainers." These local trainers then train the next cohort of providers within their organization ("Generation 2 providers").

The Train-the-Trainer Phase builds upon the first phase, the Implementation Phase (NCT04154631), in which implementation and effectiveness outcomes of two versions of TranS-C, Standard and Adapted are compared, with CMHC providers, who are trained by treatment experts. Adapted TranS-C is a version of TranS-C designed to improve 'fit' with the CMHC context. In the Train-the-Trainer Phase, the aim is to test implementation and effectiveness outcomes of Standard and Adapted TranS-C with CMHC providers who are trained and supervised within CMHCs (i.e., Generation 2 of TTT).

In the Implementation Phase, 10 CMHC clinic sites were cluster randomized to either Standard or Adapted TranS-C. Nine CMHCs continued participation into the Train-the-Trainer Phase. Within each CMHC site, patients are randomized to immediate TranS-C or to Usual Care followed by Delayed Treatment (UC-DT). Generation 2 patients (n=130) will be assessed pre, mid and post-treatment and at 6 month follow-up. UC Berkeley will coordinate the research, facilitate implementation, collect data, etc. Generation 2 providers (n=60), trained by local trainers within an established network of CMHCs, will implement TranS-C and will be assessed at pre and post-treatment. SA1 is to confirm that both Standard vs. Adapted TranS-C, compared to UC-DT, improve sleep and circadian functioning and reduce functional impairment and disorder-focused psychiatric symptoms for Generation 2 patients. SA2 is to evaluate the fit, to the CMHC context, of Standard vs. Adapted TranS-C via Generation 2 provider ratings of acceptability, appropriateness and feasibility. SA3 will examine if better fit, operationalized via Generation 2 provider ratings of acceptability, mediates the relationship between treatment condition and Generation 2 patient outcome. This research will determine if (1) sleep and circadian problems can be effectively addressed in SMI by CMHC providers trained and supervised within CMHCs via the train-the-trainer approach, (2) test two variations of TranS-C that each have unique advantages and focus on community providers and typical community patients.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the CMHC local trainers are:

* Employed in participating CMHCs
* Completed a Generation 1 TranS-C training (i.e., led by UC Berkeley expert trainers)
* Volunteer to participate and formally consent to participate

The inclusion criteria for CMHCs are:

* Publicly funded adult mental health outpatient services
* Support from CMHC leadership

The inclusion criteria for CMHC providers are:

* Employed or able to deliver client-facing services to CMHC clients
* Interest in learning and delivering TranS-C
* Volunteer to participate and formally consent to participate

Consumers must meet the following inclusion criteria:

* Aged 18 years and older
* Meet criteria for an SMI per self-report and confirmed by referring provider or administration of the Mini International Neuropsychiatric Interview (MINI) (DSM-5, Version 7.0.0) by a licensed clinical social worker on the research team
* Exhibit a sleep or circadian disturbance as determined by endorsing 4 "quite a bit" or 5 "very much" (or the equivalent for reverse scored items) on one or more PROMIS-SD questions
* Receiving the standard of care for the SMI and consent to regular communications between the research team and provider
* Consent to access their medical record and participate in assessments
* Guaranteed place to sleep for at least 2 months that is not a shelter

Exclusion Criteria:

* Presence of an active and progressive physical illness or neurological degenerative disease directly related to the onset and course of the sleep and circadian dysfunction, or making participation in the study unfeasible based on confirmation from the treating clinician and/or medical record
* Presence of substance abuse/dependence only if it makes participation in the study unfeasible
* Current active intent or plan to commit suicide (those with suicidal ideation are eligible) only if it makes participation in the study unfeasible, or homicide risk
* Night shift work >2 nights per week in the past 3 months
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (9):
- United States (9):
  - Contra Costa Health, Housing, and Homeless Services Division, Concord, California
  - Solano County Department of Health & Social Services, Behavioral Health Services, Fairfield, California
  - Kings County Behavioral Health, Hanford, California
  - Lake County Behavioral Health Services, Lucerne, California
  - Alameda County Behavioral Health Care Services, Oakland, California
  - Placer County Health and Human Services, Adult System of Care, Roseville, California
  - Monterey County Behavioral Health, Salinas, California
  - Bay Area Community Health, San Jose, California
  - County of Santa Cruz Behavioral Health Services for Children and Adults, Santa Cruz, California

REFERENCES:
- [Derived] Harvey AG, Agnew ER, Esteva Hache R, Callaway CA, Ovalle Patino E, Milner A, Spencer JM, Diaz M, Dong L, Kilbourne AM, Buysse DJ, Stice E, Sarfan LD. A randomized trial of adapted versus standard versions the transdiagnostic intervention for sleep and circadian dysfunction (TSC) implemented via facilitation and delivered by community mental health providers using train-the-trainer. Implement Sci. 2025 Nov 29;21(1):5. doi: 10.1186/s13012-025-01467-y. PMID 41318500
- [Derived] Horwitz TB, Sarfan LD, Milner AE, Varghese J, Callaway CA, Harvey AG. The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TSC) in Community Mental Health: Evaluating Self-Reported Psychiatric Disorders as a Predictor of Symptoms and Treatment Outcome. Res Sq [Preprint]. 2025 Aug 6:rs.3.rs-7189279. doi: 10.21203/rs.3.rs-7189279/v1. PMID 40799745
- [Derived] Harvey A, Agnew ER, Hache RE, Callaway CA, Patino EO, Milner A, Spencer JM, Diaz M, Dong L, Kilbourne AM, Buysse DJ, Stice E, Sarfan LD. A randomized trial of Adapted versus Standard versions the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TSC) implemented via facilitation and delivered by community mental health providers using train-the-trainer. Res Sq [Preprint]. 2025 Jul 14:rs.3.rs-6414484. doi: 10.21203/rs.3.rs-6414484/v1. PMID 40709255
- [Derived] Callaway CA, Sarfan LD, Agnew ER, Dong L, Spencer JM, Hache RE, Diaz M, Howlett SA, Fisher KR, Yates HEH, Stice E, Kilbourne AM, Buysse DJ, Harvey AG. The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) for serious mental illness in community mental health part 2: study protocol for a hybrid type 2 effectiveness-implementation cluster-randomized trial using train-the-trainer. Trials. 2023 Aug 7;24(1):503. doi: 10.1186/s13063-023-07523-6. PMID 37550730
- [Derived] Callaway CA, Sarfan LD, Agnew ER, Dong L, Spencer JM, Hache RE, Diaz M, Howlett SA, Fisher KR, Yates HEH, Stice E, Kilbourne AM, Buysse DJ, Harvey AG. The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) for serious mental illness in community mental health part 2: Study protocol for a hybrid type 2 effectiveness-implementation cluster- randomized trial using train-the-trainer. Res Sq [Preprint]. 2023 Jun 17:rs.3.rs-2943787. doi: 10.21203/rs.3.rs-2943787/v1. PMID 37398014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: CMHCs (the units) were randomized to "Standard TranS-C" or "Adapted TranS-C" but CMHCs were not further randomized to UC-DT or Immediate TranS-C. Patients within a CMHC were randomized to UC-DT or immediate TranS-C. Therefore, only "Standard TranS-C" and "Adapted TranS-C" are reported in the participant flow so that units (i.e., CMHCS) are not counted more than once across a row.
Units Other Than Participants: CMHC Sites
Groups:
- Adapted TranS-C: Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C): The Adapted version was derived from Standard TranS-C. It was developed to improve the fit of the treatment with the Community Mental Health Center (CMHC) context.
Period: Overall Study
Arm/Group | Standard TranS-C | Adapted TranS-C
Started | 22; 3 CMHC Sites | 174; 5 CMHC Sites
Providers (Providers treated patients who were in both immediate TranS-C and delayed TranS-C conditions. To increase the sample for generation 2 providers, data for all providers were analyzed (combining across UC-DT and immediate patients that they treated).) | 6; 3 CMHC Sites | 47; 5 CMHC Sites
Patients - Immediate | 8; 3 CMHC Sites | 70; 5 CMHC Sites
Patients - UC-DT (6-month follow up was collected for immediate TranS-C only. Following usual care (UC) participants in the Adapted TranS-C condition started TranS-C 4 weeks after UC, and participants in the Standard TranS-C condition started TranS-C 8 weeks after UC.) | 8; 3 CMHC Sites | 57; 5 CMHC Sites
Completed | 10; 3 CMHC Sites | 110; 5 CMHC Sites
Not Completed | 12; 0 CMHC Sites | 64; 0 CMHC Sites
Not completed — Patients lost to post or 6-month follow-up | 12 | 64

BASELINE CHARACTERISTICS:
Population: Providers treated patients who were in both immediate TranS-C and delayed TranS-C conditions. To increase the sample for generation 2 providers, data for all providers were analyzed (combining across UC-DT and immediate patients that they treated
Groups:
- Standard TranS-C (Immediate): Standard Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C): TranS-C is a psychosocial treatment designed to improve sleep and circadian functioning. It is a modular, psychosocial, skills-based approach. In this study, two version of TranS-C will be tested: Standard and Adapted.
  Standard TranS-C is modularized and delivered across eight 50-minute, weekly, individual sessions. It is comprised of 4 cross-cutting interventions featured in every session; 4 core modules that apply to the vast majority of patients; and 7 optional modules used less commonly, depending on the presentation.
  Participants in this group received Standard TranS-C immediately.
- Adapted TranS-C (Immediate): Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C): The Adapted version was derived from Standard TranS-C. It was developed to improve the fit of the treatment with the CMHC context.
  The process for developing Adapted TranS-C has been iterative and grounded in theory, data and stakeholder feedback. The core elements of the evidence-based theory of change underpinning TranS-C have been retained. Adapted TranS-C is delivered in four 20-minute, weekly, individual sessions.
  Participants in this group received Adapted TranS-C immediately.
- Standard TranS-C (UC-DT): Usual Care Delayed Treatment. Usual care in the partner CMHCs starts with a case manager who co-ordinates care and refers each client for a medication review and to various rehabilitation programs (e.g., health care, housing, nutrition, finding a job, peer monitoring).
  Participants in this group received usual care followed by delayed treatment with Standard TranS-C.
- Adapted TranS-C (UC-DT): Usual Care Delayed Treatment. Usual care in the partner CMHCs starts with a case manager who co-ordinates care and refers each client for a medication review and to various rehabilitation programs (e.g., health care, housing, nutrition, finding a job, peer monitoring).
  Participants in this group received usual care followed by delayed treatment with Adapted TranS-C.
- Standard TranS-C - Providers: Standard TranS-C is modularized and delivered across eight 50-minute, weekly, individual sessions. It is comprised of 4 cross-cutting interventions featured in every session; 4 core modules that apply to the vast majority of patients; and 7 optional modules used less commonly, depending on the presentation.
  These data reflect the characteristics of providers who delivered Standard TranS-C.
- Adapted TranS-C - Providers: The process for developing Adapted TranS-C has been iterative and grounded in theory, data and stakeholder feedback. The core elements of the evidence-based theory of change underpinning TranS-C have been retained. Adapted TranS-C is delivered in four 20-minute, weekly, individual sessions.
  These data reflect the characteristics of providers who delivered Adapted TranS-C.
- Total: Total of all reporting groups
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Standard TranS-C - Providers | Adapted TranS-C - Providers | Total
Number analyzed (Participants) | 8 | 70 | 8 | 57 | 6 | 47 | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age for patients
  Years
    number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    (all) | 43.75 (13.18) | 43.26 (15.35) | 46.25 (8.21) | 43.43 (14.43) |  |  | 43.52 (13.72)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age for providers. Population: Data not collected for this Baseline Measure from patients.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    (all) |  |  |  |  | 39.50 (12.40) | 40.21 (10.19) | 40.13 (10.33)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5 | 42 | 4 | 39 | 5 | 33 | 128
  Male | 3 | 28 | 4 | 18 | 0 | 2 | 55
  Missing/declined to answer | 0 | 0 | 0 | 0 | 1 | 12 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 18 | 1 | 8 | 1 | 8 | 40
  Not Hispanic or Latino | 4 | 52 | 6 | 49 | 4 | 25 | 140
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 14 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 5 | 0 | 2 | 0 | 0 | 7
  Asian | 0 | 0 | 0 | 3 | 1 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 6 | 2 | 7 | 0 | 0 | 15
  Black or African American | 3 | 12 | 2 | 12 | 2 | 1 | 32
  White | 2 | 32 | 2 | 22 | 1 | 24 | 83
  More than one race | 0 | 12 | 1 | 8 | 1 | 1 | 23
  Unknown or Not Reported | 3 | 3 | 1 | 3 | 1 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 8 | 70 | 8 | 57 | 6 | 47 | 196
Education [Count of Participants; unit: Participants] — Population: Data not collected for this Baseline Measure from providers.
  Participants
    number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    High school graduate or below | 3 | 6 | 0 | 5 |  |  | 14
    Some or completed college or vocational school | 4 | 45 | 4 | 34 |  |  | 87
    Some or completed graduate school | 1 | 17 | 3 | 17 |  |  | 38
    Other/ category not listed | 0 | 0 | 1 | 0 |  |  | 1
    Missing/ declined to answer | 0 | 2 | 0 | 1 |  |  | 3
Employment [Count of Participants; unit: Participants] — Population: Data not collected for this Baseline Measure from providers.
  Participants
    number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Full-time | 1 | 13 | 3 | 11 |  |  | 28
    Part-time | 2 | 10 | 1 | 9 |  |  | 22
    Not employed | 5 | 45 | 2 | 34 |  |  | 86
    Other/ category not listed | 0 | 2 | 2 | 3 |  |  | 7
Civil Status [Count of Participants; unit: Participants] — Population: Data not collected for this Baseline Measure from providers.
  Participants
    number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Partnered | 1 | 16 | 2 | 9 |  |  | 28
    Unpartnered | 7 | 54 | 5 | 47 |  |  | 113
    Other/ category not listed | 0 | 0 | 1 | 0 |  |  | 1
    Missing/ declined to answer | 0 | 0 | 0 | 1 |  |  | 1
Living Arrangement [Count of Participants; unit: Participants] — Population: Data not collected for this Baseline Measure from providers.
  Participants
    number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Alone | 2 | 14 | 0 | 11 |  |  | 27
    With family | 5 | 38 | 7 | 31 |  |  | 81
    With friend or roommate or With friend or roommate or pet | 1 | 13 | 1 | 7 |  |  | 22
    Supportive housing | 0 | 4 | 0 | 6 |  |  | 10
    Other/ category not listed | 0 | 1 | 0 | 2 |  |  | 3
    Missing/ declined to answer | 0 | 0 | 0 | 0 |  |  | 0
Government Assistance [Count of Participants; unit: Participants] — Some patients endorsed more than one government assistance category. Population: Data not collected for this Baseline Measure from providers.
  Participants
    Unemployment: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Unemployment | 0 | 2 | 0 | 1 |  |  | 3
    Medicare: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Medicare | 1 | 8 | 0 | 3 |  |  | 12
    Medicaid: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Medicaid | 2 | 26 | 2 | 20 |  |  | 50
    Social Security: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Social Security | 3 | 6 | 0 | 7 |  |  | 16
    Food Stamps: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Food Stamps | 2 | 14 | 1 | 13 |  |  | 30
    Supplemental Security Income/ Social Security Disability Insurance: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Supplemental Security Income/ Social Security Disability Insurance | 2 | 15 | 0 | 10 |  |  | 27
    Supplemental Nutrition Assistance Program: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Supplemental Nutrition Assistance Program | 1 | 8 | 0 | 6 |  |  | 15
    Other/category not listed: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Other/category not listed | 3 | 10 | 1 | 7 |  |  | 21
    Missing/declined to answer: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Missing/declined to answer | 1 | 21 | 4 | 17 |  |  | 43
Annual Household Income [Count of Participants; unit: Participants] — Population: Data not collected for this Baseline Measure from providers.
  Participants
    number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    <$10,000 | 1 | 7 | 0 | 13 |  |  | 21
    $10,000-$20,000 | 3 | 14 | 1 | 9 |  |  | 27
    $20,000-$30,000 | 3 | 6 | 2 | 4 |  |  | 15
    $30,000-$40,000 | 0 | 5 | 0 | 2 |  |  | 7
    $40,000-$50,000 | 1 | 4 | 1 | 1 |  |  | 7
    >= $50,000 | 0 | 14 | 1 | 17 |  |  | 32
    I don't know my income | 0 | 18 | 3 | 11 |  |  | 32
    Missing/ declined to answer | 0 | 2 | 0 | 0 |  |  | 2
Self-reported Diagnosis [Count of Participants; unit: Participants] — Some patients endorsed more than one self-reported diagnosis. Population: Data not collected for this Baseline Measure from providers.
  Participants
    Neurodevelopmental disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Neurodevelopmental disorders | 1 | 10 | 0 | 11 |  |  | 22
    Psychosis: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Psychosis | 3 | 20 | 0 | 13 |  |  | 36
    Bipolar Disorder: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Bipolar Disorder | 1 | 15 | 1 | 8 |  |  | 25
    Major Depressive Disorder: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Major Depressive Disorder | 4 | 31 | 3 | 28 |  |  | 66
    Anxiety disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Anxiety disorders | 3 | 30 | 5 | 34 |  |  | 72
    Obsessive- compulsive and related disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Obsessive- compulsive and related disorders | 0 | 3 | 0 | 2 |  |  | 5
    Trauma and stressor-related disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Trauma and stressor-related disorders | 1 | 14 | 1 | 17 |  |  | 33
    Dissociative disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Dissociative disorders | 0 | 0 | 0 | 0 |  |  | 0
    Personality disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Personality disorders | 0 | 2 | 0 | 0 |  |  | 2
    Feeding and eating disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Feeding and eating disorders | 0 | 0 | 0 | 0 |  |  | 0
    Substance-related and addictive disorders: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Substance-related and addictive disorders | 0 | 3 | 0 | 2 |  |  | 5
    Other/category not listed: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Other/category not listed | 0 | 1 | 2 | 0 |  |  | 3
    Missing/declined to answer: number analyzed (Participants) | 8 | 70 | 8 | 57 | 0 | 0 | 143
    Missing/declined to answer | 1 | 7 | 0 | 7 |  |  | 15
Degree Type [Count of Participants; unit: Participants] — Some providers endorsed more than one degree type. Population: Data not collected for this Baseline Measure from patients.
  Participants
    Marriage and Family Therapy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Marriage and Family Therapy |  |  |  |  | 0 | 4 | 4
    Psychology: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Psychology |  |  |  |  | 1 | 4 | 5
    Social Work: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Social Work |  |  |  |  | 4 | 15 | 19
    Nursing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Nursing |  |  |  |  | 0 | 8 | 8
    Medical: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Medical |  |  |  |  | 0 | 1 | 1
    Other/category not listed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Other/category not listed |  |  |  |  | 0 | 4 | 4
    Missing/declined to answer: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Missing/declined to answer |  |  |  |  | 1 | 12 | 13
Therapeutic Approach [Count of Participants; unit: Participants] — Some providers endorsed more than one therapeutic approach. Population: Data not collected for this Baseline Measure from patients.
  Participants
    Client Centered: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Client Centered |  |  |  |  | 5 | 29 | 34
    Family Systems: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Family Systems |  |  |  |  | 0 | 8 | 8
    Cognitive Behavioral Therapy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Cognitive Behavioral Therapy |  |  |  |  | 2 | 20 | 22
    Psychodynamic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Psychodynamic |  |  |  |  | 1 | 11 | 12
    Humanistic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Humanistic |  |  |  |  | 1 | 7 | 8
    Integrative/Holistic: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Integrative/Holistic |  |  |  |  | 0 | 2 | 2
    Missing/declined to answer: number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Missing/declined to answer |  |  |  |  | 1 | 13 | 14
Licensure [Count of Participants; unit: Participants] — Population: Data not collected for this Baseline Measure from patients.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    Licensed |  |  |  |  | 3 | 24 | 27
    Not Licensed |  |  |  |  | 2 | 11 | 13
    Missing/ declined to answer |  |  |  |  | 1 | 12 | 13
Caseload [Mean (Standard Deviation); unit: Number of patients] — Population: Data not collected for this Baseline Measure from patients.
  Number of patients
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    (all) |  |  |  |  | 33.00 (37.24) | 33.29 (40.18) | 33.26 (39.17)
Employment Duration [Mean (Standard Deviation); unit: Years] — Population: Data not collected for this Baseline Measure from patients.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    (all) |  |  |  |  | 1.20 (1.10) | 5.41 (6.23) | 4.86 (5.98)
Years Since Degree Earned [Mean (Standard Deviation); unit: Years] — Population: Data not collected for this Baseline Measure from patients.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 47 | 53
    (all) |  |  |  |  | 6.40 (6.43) | 9.63 (9.69) | 9.26 (9.39)

OUTCOME MEASURES:

1. Primary Outcome: Patient-level Outcome: Patient-Reported Outcomes Measurement Information System - Sleep DisturbanceMeasurement Information System - Sleep Disturbance
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Scale. The 8-item short version scale assesses perceived sleep problems (e.g., sleep quality, perception of sleep difficulties) over a 7-day period. Items are rated on a 5-point scale ranging from 1 (not at all) to 5 (very much). Raw scores are summed to produce a single score, resulting in a range from 8 to 40. Raw scores are converted to t-scores using treatment manuals. T-scores range from 30.5 to 77.5. A T-score of 50 indicates the population mean with a standard deviation of 10. Higher scores indicate worse sleep disturbance.
Time Frame: Baseline, mid-treatment (2/4 weeks post-baseline), post-treatment (4/8 weeks post-baseline - the UC-DT post-assessment follows the same timeframe post-usual care and delayed treatment) for Adapted/Standard TranS-C, respectively, and 6-month follow-up.
Population: Mid-treatment and 6-month follow-up assessments were collected following TranS-C but were not collected following Usual Care (UC-DT). To increase the sample size, analyses comparing Standard vs. Adapted TranS-C collapsed over immediate and UC-DT conditions (using the assessments collected after the UC-DT group started TranS-C at mid-treatment, post-treatment, and 6-month follow-up). An additional analysis also collapsed across all conditions.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Immediate TranS-C: Standard and Adapted TranS-C combined for participants randomized to the immediate condition.
- UC-DT: Standard and Adapted TranS-C combined for participants randomized to the UC-DT condition.
- Standard TranS-C: Standard Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C): TranS-C is a psychosocial treatment designed to improve sleep and circadian functioning. It is a modular, psychosocial, skills-based approach. In this study, two version of TranS-C will be tested: Standard and Adapted.
  Standard TranS-C is modularized and delivered across eight 50-minute, weekly, individual sessions. It is comprised of 4 cross-cutting interventions featured in every session; 4 core modules that apply to the vast majority of patients; and 7 optional modules used less commonly, depending on the presentation.
  Participants in this group received Standard TranS-C immediately or after usual-care delayed treatment.
- Adapted TranS-C: Adapted Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C): The Adapted version was derived from Standard TranS-C. It was developed to improve the fit of the treatment with the CMHC context.
  The process for developing Adapted TranS-C has been iterative and grounded in theory, data and stakeholder feedback. The core elements of the evidence-based theory of change underpinning TranS-C have been retained. Adapted TranS-C is delivered in four 20-minute, weekly, individual sessions.
  Participants in this group received Adapted TranS-C immediately or after usual-care delayed treatment.
- TranS-C: Collapsed across TranS-C condition (Standard, Adapted) and treatment condition (Immediate, UC-DT)
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Immediate TranS-C | UC-DT | Standard TranS-C | Adapted TranS-C | TranS-C
Number analyzed (Participants) | 8 | 70 | 8 | 57 | 78 | 65 | 16 | 127 | 143
T-score
  Baseline | 66.67 (6.44) | 62.21 (7.73) | 60.54 (5.63) | 62.24 (7.34) | 62.71 (7.69) | 62.05 (7.14) | 63.81 (6.66) | 62.23 (7.52) | 62.40 (7.42)
  Mid-treatment: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  Mid-treatment | 49.55 (2.33) | 53.81 (9.58) |  |  | 53.60 (9.39) |  | 50.08 (2.65) | 55.10 (9.27) | 54.80 (9.08)
  Post-treatment | 51.05 (15.23) | 55.06 (10.76) | 61.48 (10.37) | 61.04 (8.52) | 54.74 (11.04) | 61.08 (8.59) | 54.21 (12.22) | 55.21 (11.18) | 55.12 (11.19)
  6-month follow-up: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  6-month follow-up | 52.35 (5.83) | 52.48 (10.34) |  |  | 52.47 (10.07) |  | 54.86 (6.74) | 53.54 (10.05) | 53.63 (9.84)
Statistical Analysis 1: Comparison: Immediate TranS-C vs UC-DT; Immediate TranS-C (Standard/Adapted combined) versus UC-DT on change in sleep disturbance from pre to post; Test type: Superiority; p < 0.001, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = -7.16
Statistical Analysis 2: Comparison: Standard TranS-C vs Adapted TranS-C; Test type: Superiority; p = 0.52, Intent-to-treat, multilevel modeling — Standard TranS-C versus Adapted TranS-C on change in sleep disturbance from pre to post; Time by treatment interaction coeff. = 2.22
Statistical Analysis 3: Comparison: TranS-C; Acceptability of intervention measure (AIM) predicting sleep disturbance; Test type: Superiority; p = 0.02, Regression, Linear; Coefficient = -10.89
Statistical Analysis 4: Comparison: TranS-C; Appropriateness of intervention measure (IAM) predicting sleep disturbance; Test type: Superiority; p = 0.04, Regression, Linear; Coefficient = -6.26
Statistical Analysis 5: Comparison: TranS-C; Feasibility of intervention measure (FIM) predicting sleep disturbance; Test type: Superiority; p = 0.001, Regression, Linear; Coefficient = -10.37

2. Primary Outcome: Provider-level Outcome: Acceptability Intervention Measure
Description: Assesses provider perceptions of the acceptability of the treatment intervention using a self-report questionnaire. The 4-item scale is rated on a 5-point scale from 1 (completely disagree) to 5 (completely agree). A total score is calculated by averaging all four items. Total scores range from 1 to 5, with higher scores indicating greater perceptions of acceptability.
Time Frame: Baseline, mid-treatment (2 weeks post-baseline for Adapted TranS-C and 4 weeks post-baseline for Standard TranS- C), post-treatment (4 weeks post-baseline for Adapted TranS-C and 8 weeks post-baseline for Standard TranS-C).
Population: Acceptability Intervention Measure was collected only from providers. To increase the sample size, and because providers treated patients who could have been in either the immediate or UC-DT conditions, we analyzed by collapsing across immediate and UC-DT for providers. For some analyses, data were collapsed across Standard and Adapted TranS-C. This measure was not assessed following usual care.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard TranS-C - Providers: Standard TranS-C is modularized and delivered across eight 50-minute, weekly, individual sessions. It is comprised of 4 cross-cutting interventions featured in every session; 4 core modules that apply to the vast majority of patients; and 7 optional modules used less commonly, depending on the presentation.
- Adapted TranS-C - Providers: The process for developing Adapted TranS-C has been iterative and grounded in theory, data and stakeholder feedback. The core elements of the evidence-based theory of change underpinning TranS-C have been retained. Adapted TranS-C is delivered in four 20-minute, weekly, individual sessions.
- TranS-C - Providers: Collapsed across Standard and Adapted TranS-C.
Arm/Group | Standard TranS-C - Providers | Adapted TranS-C - Providers | TranS-C - Providers
Number analyzed (Participants) | 6 | 47 | 53
score on a scale
  Baseline | 4.90 (0.22) | 4.74 (0.41) | 4.76 (0.39)
  Mid-treatment | 5.00 (0.00) | 4.64 (0.44) | 4.65 (0.44)
  Post-treatment | 5.00 (0.00) | 4.54 (0.58) | 4.56 (0.57)

3. Secondary Outcome: Patient-level Outcome: Patient-Reported Outcomes Measurement Information System - Sleep Related Impairment
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Impairment Scale. The 8-item short version scale assesses perceived sleep problems during waking hours (e.g., alertness, sleepiness, tiredness) over a 7-day period. Items are rated on a 5-point scale ranging from 1 (not at all) to 5 (very much). Raw scores are summed to produce a single score, resulting in a range from 8 to 40. Raw scores are converted to t-scores using treatment manuals. T-scores range from 30.1 to 80.1. A T-score of 50 indicates the population mean with a standard deviation of 10. Higher scores indicate worse sleep-related impairment.
Time Frame: as for outcome 1
Population: Mid-treatment and 6-month follow-up assessments were collected following TranS-C but were not collected following Usual Care (UC-DT). To increase the sample size, analyses comparing Standard vs. Adapted TranS-C collapsed over immediate and UC-DT conditions (using the assessments collected post TranS-C for the UC-DT group). An additional analysis also collapsed across all conditions.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Immediate TranS-C | UC-DT | Standard TranS-C | Adapted TranS-C | TranS-C
Number analyzed (Participants) | 8 | 70 | 8 | 57 | 78 | 65 | 16 | 127 | 143
T-score
  Baseline | 63.12 (10.63) | 60.30 (8.57) | 59.24 (10.79) | 60.09 (8.58) | 60.59 (8.76) | 59.98 (8.79) | 61.18 (10.54) | 60.20 (8.54) | 60.31 (8.75)
  Mid-treatment: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  Mid-treatment | 60.20 (5.80) | 55.67 (10.66) |  |  | 55.89 (10.47) |  | 55.83 (8.82) | 56.76 (10.45) | 56.70 (10.30)
  Post-treatment | 48.65 (12.87) | 52.80 (11.90) | 59.66 (6.61) | 57.71 (8.58) | 52.46 (11.90) | 57.88 (8.39) | 52.74 (10.56) | 53.54 (11.14) | 53.48 (11.03)
  6-month follow-up: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  6-month follow-up | 50.75 (9.05) | 53.82 (11.29) |  |  | 53.62 (11.12) |  | 54.27 (9.82) | 54.71 (10.90) | 54.68 (10.79)
Statistical Analysis 1: Comparison: Immediate TranS-C vs UC-DT; Treatment condition (Standard/Adapted TranS-C versus UC-DT) on change in sleep- related impairment from pre to post; Test type: Superiority; p = 0.001, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = -6.44
Statistical Analysis 2: Comparison: Standard TranS-C vs Adapted TranS-C; Standard TranS-C versus Adapted TranS-C on change in sleep-related impairment from pre to post; Test type: Superiority; p = 0.72, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = 1.36
Statistical Analysis 3: Comparison: TranS-C; Acceptability of intervention measure (AIM) predicting sleep-related impairment; Test type: Superiority; p = 0.30, Regression, Linear; Coefficient = -3.90
Statistical Analysis 4: Comparison: TranS-C; Appropriateness of intervention measure (IAM) predicting sleep-related impairment; Test type: Superiority; p = 0.78, Regression, Linear; Coefficient = 0.79
Statistical Analysis 5: Comparison: TranS-C; Feasibility of intervention measure (FIM) predicting sleep-related impairment; Test type: Superiority; p = 0.15, Regression, Linear; Coefficient = -4.45

4. Secondary Outcome: Patient-level Outcome: Composite Sleep Health Score
Description: Composite Sleep Health Score is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint sleep fluctuation across a 7-day sleep diary < 1 hour), Satisfaction (Sleep quality question on PROMIS-Sleep Disturbance (PROMIS = Patient-Reported Outcomes Measurement Information System)), Alertness (Daytime sleepiness question on PROMIS-Sleep Related Impairment (PROMIS = Patient-Reported Outcomes Measurement Information System)), Timing (Mean midpoint sleep across the 7 day sleep diary between 2 and 4 AM), Efficiency (Average sleep efficiency based on the 7 day sleep diary ≥ 85%), and Duration (Total Sleep Time average based on 7 day sleep diary between 7 and 9 hours). Each dimension was dichotomized such that 1 = good /yes; 0 = poor/no). Total composite sleep health score ranges from 0 to 6, with larger values indicating better sleep health.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Immediate TranS-C | UC-DT | Standard TranS-C | Adapted TranS-C | TranS-C
Number analyzed (Participants) | 8 | 70 | 8 | 57 | 78 | 65 | 16 | 127 | 143
score on a scale
  Baseline | 3.00 (1.10) | 2.25 (1.29) | 2.29 (1.50) | 2.45 (1.47) | 2.31 (1.28) | 2.43 (1.46) | 2.62 (1.33) | 2.33 (1.37) | 2.36 (1.36)
  Mid-treatment: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  Mid-treatment | 3.50 (2.12) | 3.28 (1.54) |  |  | 3.29 (1.54) |  | 3.50 (1.73) | 3.05 (1.54) | 3.08 (1.55)
  Post-treatment | 3.33 (2.52) | 3.07 (1.59) | 3.00 (1.41) | 2.66 (1.45) | 3.09 (1.63) | 2.69 (1.44) | 2.50 (2.07) | 3.07 (1.52) | 3.03 (1.56)
  6-month follow-up: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  6-month follow-up | 4.00 (1.41) | 2.94 (1.62) |  |  | 3.02 (1.62) |  | 3.57 (1.62) | 2.90 (1.52) | 2.95 (1.53)
Statistical Analysis 1: Comparison: Immediate TranS-C vs UC-DT; Treatment condition (Standard/Adapted TranS-C versus UC-DT) on change in Composite Sleep Health Score from pre to post; Test type: Superiority; p = 0.09, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = 0.55
Statistical Analysis 2: Comparison: Standard TranS-C vs Adapted TranS-C; Standard TranS-C versus Adapted TranS-C on change in sleep health from pre to post; Test type: Superiority; p = 0.11, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = 1.05
Statistical Analysis 3: Comparison: TranS-C; Acceptability of intervention measure (AIM) predicting sleep health; Test type: Superiority; p = 0.59, Regression, Linear; Coefficient = 0.45
Statistical Analysis 4: Comparison: TranS-C; Appropriateness of intervention measure (IAM) predicting sleep health; Test type: Superiority; p = 0.14, Regression, Linear; Coefficient = 0.72
Statistical Analysis 5: Comparison: TranS-C; Feasibility of intervention measure (FIM) predicting sleep health; Test type: Superiority; p = 0.06, Regression, Linear; Coefficient = 0.89

5. Secondary Outcome: Patient-level Outcome: Sheehan Disability Scale
Description: The Sheehan Disability Scale (SDS) assesses impairment in work/school, social, and family life. Items are rated on a scale from 0 (not at all) to 10 (extremely). Items are summed to produce a single score. Scores range from 0 to 30, with higher scores indicating higher functional impairment.
Time Frame: Baseline, post-treatment (4/8 weeks post-baseline - the UC-DT post-assessment follows the same timeframe post-usual care and delayed treatment) for Adapted/Standard TranS-C, respectively, and 6-month follow-up.
Population: 6-month follow-up assessments were collected following TranS-C but were not collected following Usual Care (UC-DT). To increase the sample size, analyses comparing Standard vs. Adapted TranS-C collapsed over immediate and UC-DT conditions (using the assessments collected after the UC-DT group started TranS-C at post-treatment, and 6-month follow-up). An additional analysis also collapsed across all conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Immediate TranS-C | UC-DT | Standard TranS-C | Adapted TranS-C | TranS-C
Number analyzed (Participants) | 8 | 70 | 8 | 57 | 78 | 65 | 16 | 127 | 143
score on a scale
  Baseline | 15.25 (6.63) | 12.49 (7.72) | 11.75 (10.07) | 11.88 (7.04) | 12.77 (7.62) | 11.86 (7.38) | 13.50 (8.43) | 12.21 (7.40) | 12.36 (7.50)
  Post-treatment | 6.50 (6.35) | 7.98 (7.06) | 10.80 (7.66) | 11.10 (7.51) | 7.86 (6.95) | 11.07 (7.46) | 8.86 (7.73) | 8.36 (6.47) | 8.40 (6.54)
  6-month follow-up: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  6-month follow-up | 9.75 (8.26) | 8.51 (7.06) |  |  | 8.59 (7.07) |  | 9.71 (8.46) | 8.70 (7.05) | 8.77 (7.11)
Statistical Analysis 1: Comparison: Immediate TranS-C vs UC-DT; Treatment condition (Standard/Adapted TranS-C versus UC-DT) on change in functional impairment from pre to post; Test type: Superiority; p = 0.002, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = -4.33
Statistical Analysis 2: Comparison: Immediate TranS-C vs UC-DT; Structural equation modeling (SEM) was used to test whether the relationship between TranS-C condition (Immediate vs. UC-DT) and functional impairment (Sheehan Disability Scale) at post was mediated by sleep disturbance (PROMIS-SD) at post. The parameter of interest was the indirect effect; Test type: Superiority; p = 0.002, SEM; Coefficient of indirect effect = -2.20, 95% CI 2-sided [-3.57 to -0.83]
Statistical Analysis 3: Comparison: Immediate TranS-C vs UC-DT; Structural equation modeling (SEM) was used to test whether the relationship between TranS-C condition (Immediate vs. UC-DT) and functional impairment (Sheehan Disability Scale) at post was mediated by sleep-related impairment (PROMIS-SRI). The parameter of interest was the indirect effect at post; Test type: Superiority; p = 0.001, SEM; Coefficient of indirect effect = -2.76, 95% CI 2-sided [-4.44 to -1.08]
Statistical Analysis 4: Comparison: Standard TranS-C vs Adapted TranS-C; Standard TranS-C versus Adapted TranS-C on change in functional impairment from pre to post; Test type: Superiority; p = 0.78, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = 0.84
Statistical Analysis 5: Comparison: TranS-C; Acceptability of intervention measure (AIM) predicting functional impairment; Test type: Superiority; p = 0.49, Regression, Linear; Coefficient = -1.41
Statistical Analysis 6: Comparison: TranS-C; Appropriateness of intervention measure (IAM) predicting functional impairment; Test type: Superiority; p = 0.27, Regression, Linear; Coefficient = -1.62
Statistical Analysis 7: Comparison: TranS-C; Feasibility of intervention measure (FIM) predicting functional impairment; Test type: Superiority; p = 0.09, Regression, Linear; Coefficient = -2.07

6. Secondary Outcome: Patient-level Outcome: The Diagnostic and Statistical Manual of Mental Disorders Cross-Cutting Symptom Measure
Description: The Diagnostic and Statistical Manual of Mental Disorders Cross-Cutting Symptom Measure (DSM-5) assesses psychiatric symptoms across 13 mental health domains. Participants rate on a 5-point scale how often they were bothered by each symptom on a scale from 0 (not at all) to 4 (nearly every day). Scores range from 0 to 52, with higher scores indicating more severe symptoms.
Time Frame: as for outcome 5
Population: 6-month follow-up assessments were collected following TranS-C but were not collected following Usual Care (UC-DT). To increase the sample size, analyses comparing Standard vs. Adapted TranS-C collapsed over immediate and UC-DT conditions (using the assessments collected after the UC-DT group started TranS-C at mid-treatment, post-treatment, and 6-month follow-up). An additional analysis also collapsed across all conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Immediate TranS-C | UC-DT | Standard TranS-C | Adapted TranS-C | TranS-C
Number analyzed (Participants) | 8 | 70 | 8 | 57 | 78 | 65 | 16 | 127 | 143
score on a scale
  Baseline | 25.38 (8.93) | 23.48 (8.70) | 18.75 (5.18) | 23.25 (9.48) | 22.69 (9.15) | 23.68 (8.69) | 22.06 (7.84) | 23.37 (9.03) | 23.23 (8.89)
  Post-treatment | 14.00 (10.68) | 17.91 (9.61) | 20.60 (5.32) | 20.67 (8.74) | 17.59 (9.64) | 20.67 (8.46) | 16.14 (8.07) | 18.00 (9.34) | 17.84 (9.20)
  6-month follow-up: number analyzed (Participants) | 8 | 70 | 0 | 0 | 78 | 0 | 16 | 127 | 143
  6-month follow-up | 14.25 (8.30) | 18.47 (10.16) |  |  | 18.19 (10.04) |  | 17.29 (7.20) | 18.24 (9.51) | 18.18 (9.34)
Statistical Analysis 1: Comparison: Immediate TranS-C vs UC-DT; Treatment condition (Standard/Adapted TranS-C versus UC-DT) on change in psychiatric symptoms from pre to post; Test type: Superiority; p = 0.002, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = -4.25
Statistical Analysis 2: Comparison: Immediate TranS-C vs UC-DT; Structural equation modeling (SEM) was used to test whether the relationship between TranS-C condition (Immediate vs. UC-DT) and psychiatric symptoms (Diagnostic and Statistical Manual of Mental Disorders Cross-Cutting Symptom Measure) at post was mediated by sleep disturbance (PROMIS-SD) at post. The parameter of interest was the indirect effect; Test type: Superiority; p = 0.02, SEM; Coefficient of indirect effect = -1.95, 95% CI 2-sided [-3.54 to -0.36]
Statistical Analysis 3: Comparison: Immediate TranS-C vs UC-DT; Structural equation modeling (SEM) was used to test whether the relationship between TranS-C condition (Immediate vs. UC-DT) and psychiatric symptoms (Diagnostic and Statistical Manual of Mental Disorders Cross-Cutting Symptom Measure) at post was mediated by sleep-related impairment (PROMIS-SRI) at post. The parameter of interest was the indirect effect; Test type: Superiority; p = 0.01, SEM; Coefficient of indirect effect = -1.62, 95% CI 2-sided [-2.87 to -0.38]
Statistical Analysis 4: Comparison: Standard TranS-C vs Adapted TranS-C; Standard TranS-C versus Adapted TranS-C on change in psychiatric symptoms from pre to post; Test type: Superiority; p = 0.56, Intent-to-treat, multilevel modeling; Time by treatment interaction coeff. = 1.79
Statistical Analysis 5: Comparison: TranS-C; Acceptability of intervention measure (AIM) predicting psychiatric symptoms; Test type: Superiority; p = 0.34, Regression, Linear; Coefficient = -3.46
Statistical Analysis 6: Comparison: TranS-C; Appropriateness of intervention measure (IAM) predicting psychiatric symptoms; Test type: Superiority; p = 0.01, Regression, Linear; Coefficient = -5.54
Statistical Analysis 7: Comparison: TranS-C; Feasibility of intervention measure (FIM) predicting psychiatric symptoms; Test type: Superiority; p = 0.01, Regression, Linear; Coefficient = -5.65

7. Secondary Outcome: Provider-level Outcome: Intervention Appropriateness Measure
Description: Assesses provider perceptions of the appropriateness of the treatment intervention using a self-report questionnaire. The 4-item scale is rated on a 5-point scale from 1 (completely disagree) to 5 (completely agree). A total score is calculated by averaging all four items. Total scores range from 1 to 5, with higher scores indicating greater perceptions of appropriateness.
Time Frame: as for outcome 2
Population: Intervention Appropriateness Measure was collected only from providers. To increase the sample size, and because providers treated patients who could have been in either the immediate or UC-DT conditions, we analyzed by collapsing across immediate and UC-DT for providers. For some analyses, data were collapsed across Standard and Adapted TranS-C. This measure was not assessed following usual care.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- TranS-C Providers: Collapsed across Standard and Adapted TranS-C.
Arm/Group | Standard TranS-C - Providers | Adapted TranS-C - Providers | TranS-C Providers
Number analyzed (Participants) | 6 | 47 | 53
score on a scale
  Baseline | 5.00 (0.00) | 4.79 (0.35) | 4.82 (0.33)
  Mid-treatment | 4.83 (0.29) | 4.56 (0.52) | 4.58 (0.51)
  Post-treatment | 4.75 (0.50) | 4.39 (0.67) | 4.41 (0.67)

8. Secondary Outcome: Provider-level Outcome: Feasibility of Intervention Measure
Description: Assesses provider perceptions of the feasibility of the treatment intervention using a self-report questionnaire. The 4- item scale is rated on a 5-point scale from 1 (completely disagree) to 5 (completely agree). A total score is calculated by averaging all four items. Total scores range from 1 to 5, with higher scores indicating greater perceptions of feasibility.
Time Frame: Baseline, mid-treatment (2 weeks post-baseline for Adapted TranS-C and 4 weeks post-baseline for Standard TranS-C), post-treatment (4 weeks post-baseline for Adapted TranS-C and 8 weeks post-baseline for Standard TranS-C).
Population: Feasibility of Intervention Measure was collected only from providers. To increase the sample size, and because providers treated patients who could have been in either the immediate or UC-DT conditions, we analyzed by collapsing across immediate and UC-DT for providers. For some analyses, data were collapsed across Standard and Adapted TranS-C. This measure was not assessed following usual care.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard TranS-C - Providers | Adapted TranS-C - Providers | TranS-C - Providers
Number analyzed (Participants) | 6 | 47 | 53
score on a scale
  Baseline | 4.95 (0.11) | 4.59 (0.57) | 4.64 (0.54)
  Mid-treatment | 4.83 (0.29) | 4.60 (0.54) | 4.61 (0.53)
  Post-treatment | 4.44 (0.72) | 4.42 (0.65) | 4.43 (0.65)

9. Other Pre Specified Outcome: Patient-level Outcome: Midpoint of Sleep Measure
Description: Assesses circadian functioning by calculating the midpoint between falling asleep time and rise time.
Time Frame: Change from baseline, to mid-treatment, which is 2 or 4 weeks after the beginning of treatment, to post-treatment, which is 6 or 10 weeks after the beginning of treatment, and to 6-month follow-up.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Patient-level Outcome: Alcohol Intake
Description: Assesses past 30-day quantity and frequency of alcohol intake using a self-report questionnaire.
Time Frame: Change from baseline to post-treatment, which is 6 or 10 weeks after the beginning of treatment, and to 6-month follow-up.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Patient-level Outcome: Substances Intake
Description: Assesses past 30-day frequency of substance use using a self-report questionnaire.
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patient-level Outcome: Tobacco Intake
Description: Assesses past 30-day quantity and frequency of tobacco intake using a self-report questionnaire.
Time Frame: as for outcome 10
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Patient-level Outcome: Caffeine Intake
Description: Assesses past 30-day quantity and frequency of caffeine intake using a self-report questionnaire.
Time Frame: as for outcome 10
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Patient-level Outcome: Suicidal Ideation Questionnaire
Description: Assesses past 30-day suicidal ideation using a self-report questionnaire.
Time Frame: as for outcome 10
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Patient-level Outcome: Credibility Expectancy Questionnaire
Description: Measures the credibility and expectation of improvement from TranS-C. The questionnaire includes 4 items.
Time Frame: Once at post-treatment, which is 6 or 10 weeks after the beginning of treatment.
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Patient-level Outcome: Utilization Questionnaire
Description: Measures the elements of TranS-C that are most used.
Time Frame: Once at post-treatment, which is 6 or 10 weeks after the beginning of treatment.
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Patient-level Outcome: Utilization Questionnaire
Description: Measures the elements of TranS-C that are most used.
Time Frame: Once at 6-month follow-up after treatment ends.
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Patient-level Outcome: Duke Checklist of Medical Conditions & Symptoms
Description: Assesses physical illness or neurological degenerative disease directly related to the onset and course of the sleep and circadian dysfunction.
Time Frame: Once at baseline.
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Provider-level Outcome: Checklist of Modules Delivered
Description: Assesses which treatment modules were delivered by the providers using a self-report checklist.
Time Frame: Once at each session between patient and provider.
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Provider-level Outcome: Adaptations to Evidence-Based Practices Scale
Description: Assesses ad hoc modifications the provider made to the treatment using a self-report questionnaire.
Time Frame: Once at post-treatment, which is 6 or 10 weeks after the beginning of treatment.
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Provider-level Outcome: Use of TranS-C Assessment
Description: Assesses if providers continue to use TranS-C in a self-report questionnaire.
Time Frame: Once during the 1 year sustainment phase.
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Provider-level Outcome: Session Attendance and Duration Log
Description: Collect session date and duration (length of session).
Time Frame: Once at each session between patient and provider.
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Provider-level Outcome: Training Evaluation/Knowledge Test
Description: Provider evaluation of the training; provider knowledge of content covered in the training; provider willingness and confidence in delivering TranS-C.
Time Frame: Through the first 2.5 years of the study, an average of 4 per month
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Provider-level Outcome: Gold Standard Training Elements
Description: Extent of gold standard training elements present in each training session, with respect to content and technique.
Time Frame: Through the first 2.5 years of the study, an average of 4 per month
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Provider-level Outcome: Number of TranS-C Sessions
Description: Number of sessions delivered to each enrolled patient by each provider.
Time Frame: Once per patient at posttreatment, which is 6 or 10 weeks after the beginning of treatment
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Facilitator-level Outcome: Implementation Log
Description: Weekly record of facilitator activities, amount of time per activity, county, year, type of communication, implementation strategies, target(s), intended outcome(s).
Time Frame: Up to 30 months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Facilitator-level Outcome: Meeting Log
Description: Weekly record of community meeting details as applicable, including: county, generation, level of contact (i.e., leadership, providers), type/modality of contact, length of meeting, number of attendees, recording, general description, standardized description, main presenter and role of UC Berkeley staff.
Time Frame: Up to 30 months
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Patient-level Outcome: Patient-Reported Outcomes Measurement Information System - Sleep Disturbance
Description: Assesses perceived functional impairments related to sleep problems using a self-report questionnaire. The minimum value is 8. The maximum value is 40. Higher scores mean more sleep disturbance (worse outcome).
Time Frame: Change from baseline to mid-treatment, which is 2 or 4 weeks after the beginning of treatment
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Provider-level Outcome: Acceptability Intervention Measure
Description: Assesses provider perceptions of the appropriateness of the treatment intervention using a self-report questionnaire and provider feedback.
Time Frame: Change from baseline to mid-treatment, which is 2 or 4 weeks after the beginning of treatment for each client
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 months.
Description: Providers treated patients who could have been in either the immediate or UC-DT conditions. Therefore, we analyzed by collapsing across immediate and UC-DT for providers.
Arm/Group | Standard TranS-C (Immediate) | Adapted TranS-C (Immediate) | Standard TranS-C (UC-DT) | Adapted TranS-C (UC-DT) | Standard TranS-C - Providers | Adapted TranS-C - Providers
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/70 | 0/8 | 0/57 | 0/6 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/70 | 0/8 | 0/57 | 0/6 | 0/47
Other Adverse Events (participants affected / at risk) | 0/8 | 0/70 | 0/8 | 0/57 | 0/6 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT05805657/Prot_SAP_000.pdf